CLINICAL TRIAL: NCT02059265
Title: A Phase II Trial of DCTD-Sponsored Dasatinib in Recurrent/Persistent Ovary, Fallopian Tube, Primary Peritoneal, and Endometrial Clear Cell Carcinoma Characterized for the Retention or Loss of BAF250a Expression
Brief Title: Dasatinib in Treating Patients With Recurrent or Persistent Ovarian, Fallopian Tube, Endometrial or Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim monitoring
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00209; NCI-2014-00209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0283; GOG-0283 (Other: NRG Oncology); GOG-0283 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Clear Cell Adenocarcinoma; Ovarian Clear Cell Cystadenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well dasatinib works in treating patients with ovarian, fallopian tube, endometrial, or peritoneal cancer that has come back or is persistent. Dasatinib may shrink patients' tumors by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical activity of dasatinib in patients with recurrent or persistent ovarian, fallopian tube, primary peritoneal, and endometrial clear cell carcinoma using objective tumor response (complete and partial): in patients without loss of BRG-associated factor 250a (BAF250a) expression and in patients with loss of BAF250a expression.

SECONDARY OBJECTIVES:

I. To examine the nature and degree of toxicity in this patient population treated with this regimen in patients with and without loss of BAF250a expression.

II. To examine the progression-free survival and overall survival for this patient population receiving dasatinib in patients with and without loss of BAF250a expression.

TERTIARY OBJECTIVES:

I. To examine the agreement between BAF250a immunohistochemistry and AT rich interactive domain 1A (SWI-like) (ARID1A) mutation status using next generation sequencing performed in formalin-fixed, paraffin-embedded tumor tissue.

OUTLINE:

Patients receive dasatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent ovarian, fallopian tube, peritoneum, and endometrial clear cell carcinoma; primary tumors must be at least 50% clear cell histomorphology in order to be eligible or have a histologically documented recurrence with at least 50% clear cell histomorphology; in addition, the tumors should be negative for expression of Wilms tumor 1 (WT-1) antigen (with the exception of endometrial cancers where WT-1 stains are not required) and estrogen receptor (ER) antigen by immunohistochemistry; focal, weak, ER staining of tumor cells (< 5%) is permitted; appropriate tissue sections must be available for histologic evaluation for central pathology review by Gynecologic Oncology Group (GOG); immunohistochemical stained slides for ER and WT-1 antigen must be available for review by GOG

  * If the primary tumor had at least 50% clear cell histomorphology, a biopsy of the recurrent or persistent tumor is not required; however, immunohistochemical studies of the primary tumor for ER and WT-1 antigens should be performed and the slides submitted to the GOG for review; the percentage of clear cell histomorphology must be documented in the pathology report or in an addendum to the original report; if slides of the primary tumor are not available for review due to disposal of slides by the histology laboratory (typically 10 years after diagnosis), biopsy of recurrent or persistent disease is required
  * If the primary tumor had less than 50% clear cell histomorphology (or if slides of the primary tumor are not available for review), a biopsy of the recurrent or persistent tumor is required to confirm at least 50% clear cell histomorphology and lack of immuno-reactivity for ER and WT-1 antigens by immunohistochemistry; the percentage of involvement must be documented in the pathology report or in an addendum to the original report
* Patients must have results from the determination of BAF250a immunohistochemistry (IHC) status and must have a BAF250a expression status that is currently open to enrollment
* All patients must have measurable disease; measurable disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1); measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography [CT], magnetic resonance imaging [MRI] or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease; patients are allowed to receive, but are not required to receive, two additional cytotoxic regimens for management of recurrent or persistent disease
* Patients must be >= 3 weeks from last chemotherapy or radiation (6 weeks for nitrosoureas or mitomycin)
* Patients must have progressed on, be ineligible for, or have declined participation in GOG-0254 provided that protocol is actively accruing patients
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Creatinine =< 1.5 times the upper limit of normal (ULN) OR creatinine clearance >= 60 mL/min/1.73 m^2
* Bilirubin =< 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase ALT (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Patients who are on concomitant medications that are STRONG inducers or inhibitors of the cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) enzyme should stop 2 weeks prior to first dose of dasatinib, if all other eligibility has been confirmed
* Corrected QT (QTc) interval on electrocardiogram must be =< 480 msec (Fridericia correction)
* Patients who have received one prior regimen must have a GOG performance status of 0, 1 or 2; patients who have received two or more prior regimens must have GOG performance status of 0 or 1
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Prior treatment with dasatinib, imatinib or nilotinib
* Patients with symptomatic effusions (pleural, pericardial, or peritoneal) and/or those who have required a procedure for symptomatic effusions within 4 weeks of start of dasatinib are ineligible
* Patients with a history of cardiac disease including: (1) uncontrolled angina, congestive heart failure, or myocardial infarction within six months prior to study entry, (2) congenital long QT syndrome, (3) clinical significant ventricular arrhythmias
* The concomitant use of histamine (H)2 blockers and proton pump inhibitors (PPIs) with dasatinib is not recommended; the use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy; if antacid therapy is needed, the antacid dose should be administered two hours before or after the dose of dasatinib; patients who cannot tolerate discontinuation of H2 blockers or PPIs are ineligible
* Therapeutic anticoagulation is not contraindicated, but for those patients on therapeutic anticoagulation, alteration in coagulation parameters is expected following initiation of dasatinib; for patients on therapeutic anticoagulation, coagulation parameters should be assessed weekly for the first cycle following initiation of dasatinib, weekly for the first cycle following a dose reduction, and weekly for a minimum of two weeks after stopping dasatinib
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Patients who are pregnant or nursing; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 3 months after completion of therapy; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a negative serum pregnancy test within 72 hours of starting drug is required
* Patients who have a major surgical procedure, or significant traumatic injury within 28 days prior to the first date of treatment on this study, or anticipation of need for major surgical procedure during the course of the study; patients with placement of vascular access device or core biopsy within 7 days prior to the first date of treatment on this study
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients who are unable to swallow pills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02-14 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Hyman, Principal Investigator — NRG Oncology
Locations (227):
- United States (227):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on 2/3/2014 and accrued 35 (28 treated and eligible) of a planned 62 patients. The study was closed on 8/10/2016, after evaluation of the stage 1 data.
Pre-assignment Details: Four patients were deemed ineligible and three patients were never treated; 28 patients were evaluable for efficacy and safety.
Period: Overall Study
Arm/Group | Treatment (Dasatinib)
Started | 32
Completed | 28
Not Completed | 4
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib: Dasatinib - 140 mg by mouth, once daily, on days 1-28 (one cycle = 28 days) until disease progression or adverse effects prohibit further therapy
Arm/Group | Dasatinib
Number analyzed (Participants) | 28
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0
  30-39 years | 2
  40-49 years | 3
  50-59 years | 10
  60-69 years | 8
  70-79 years | 4
  >= 80 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.1
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST 1.1 defines complete response as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and the disappearance of all non-target lesions and normalization of tumor marker level. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; then every 3 months x 2; then every 6 months thereafter until disease progression for up to 5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 28
Participants | 1

2. Secondary Outcome: Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 28
Months | 16.92 [4.57 to 30.52]

3. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: PFS will be characterized with Kaplan-Meier plots and estimates of the median time until death or progression.
Time Frame: Duration of time from start of treatment to time of progression or death, whichever occurs first, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 28
Months | 2.14 [1.58 to 7.29]

4. Secondary Outcome: Incidence of Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: The frequency and severity of all toxicities are tabulated.
Time Frame: Up to 5 years
Measure: Number; unit: Count of Participants with >= grade 3 AE
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 28
Count of Participants with >= grade 3 AE | 20

5. Other Pre Specified Outcome: ARID1A Mutation Status in Formalin-fixed, Paraffin Embedded Tissue Using Next-generation Exon-capture Sequencing
Description: ARID1A mutation status will be tabulated to determine the correlation between BAF250a IHC and ARID1A mutations.
Time Frame: Up to 5 years
Population: ARID1A information was available for 26 of 35 patients. Missing data is attributed to assay failure.
Measure: Number (95% Confidence Interval); unit: Spearman Correlation Coefficient
Arm/Group | Treatment (Dasatinib)
Number analyzed (Participants) | 26
Spearman Correlation Coefficient | 0.82 [0.59 to 1.00]

ADVERSE EVENTS:
Time Frame: Up to 5 Years
Arm/Group | Treatment (Dasatinib)
All-Cause Mortality (participants affected / at risk) | 24/28
Serious Adverse Events (participants affected / at risk) | 16/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Dasatinib) (N=28)
Cardiac Arrest (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Duodenal Obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Stomach Pain (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Lung Infection (Infections and infestations) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Dasatinib) (N=28)
Anemia (Blood and lymphatic system disorders) | 21
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Duodenal Obstruction (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 7
Bloating (Gastrointestinal disorders) | 3
Stomach Pain (Gastrointestinal disorders) | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 11
Mucositis Oral (Gastrointestinal disorders) | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 19
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Jejunal Obstruction (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Pain (General disorders) | 1
Flu Like Symptoms (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Edema Limbs (General disorders) | 3
Fatigue (General disorders) | 20
Fever (General disorders) | 5
Sinusitis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Abdominal Infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 1
Weight Gain (Investigations) | 1
Platelet Count Decreased (Investigations) | 3
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 2
Creatinine Increased (Investigations) | 7
Neutrophil Count Decreased (Investigations) | 3
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 6
Aspartate Aminotransferase Increased (Investigations) | 1
Alkaline Phosphatase Increased (Investigations) | 5
Alanine Aminotransferase Increased (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Tremor (Nervous system disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Urinary Urgency (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Breast Pain (Reproductive system and breast disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Thromboembolic Event (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hot Flashes (Vascular disorders) | 3
Flushing (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT02059265/Prot_SAP_000.pdf